CLINICAL TRIAL: NCT03041181
Title: Randomized Phase II Trial of Single Agent Chemotherapy Plus Nivolumab or Single Agent Chemotherapy Alone in Patients With Advanced Squamous or Non-squamous NSCLC With Primary Resistance to Prior PD-1 or PDL-1 Inhibitor
Brief Title: Single Agent Chemotherapy +/- Nivolumab in Patients With Advanced Squamous or Non-squamous NSCLC With Primary Resistance to Prior PD-1 or PDL-1 Inhibitor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder decision - lack of accrual
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Hoosier Cancer Research Network (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN15-233
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer (NSCLC); Adenocarcinoma of the Lung; Lung Cancer; Squamous Cell Lung Cancer
Keywords: Nivolumab; BMS-936558-01; Anti-PD-1 Antibody; Docetaxel; Pemetrexed; Gemcitabine
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms | interventions — Docetaxel; Nivolumab; Gemcitabine; Pemetrexed

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A - Single Agent Chemotherapy + Nivolumab (Experimental): Single Agent Chemotherapy of choice plus nivolumab:
  Taxotere Pemetrexed Gemcitabine
  Interventions: Drug: Docetaxel; Drug: Nivolumab; Drug: Gemcitabine; Drug: Pemetrexed
- Arm B - Single Agent Chemotherapy (Active Comparator): Single Agent Chemotherapy of choice Taxotere Pemetrexed Gemcitabine
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
  Other Names: Taxotere
Drug: Nivolumab — Nivolumab 360 mg IV Day 1 of each cycle (21 days = 1 cycle)
  Other Names: BMS-936558-01; Opdivo
  Arms: Arm A - Single Agent Chemotherapy + Nivolumab
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV Day 1 and Day 8 of each cycle (21 days = 1 cycle)
  Other Names: Gemzar
Drug: Pemetrexed — Pemetrexed 500 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
  Other Names: Alimta

SUMMARY:
This is a randomized phase II study assessing the activity of single agent chemotherapy combined with nivolumab (Arm A) compared to single agent chemotherapy alone (Arm B) in squamous or non-squamous NSCLC subjects with primary resistance to prior PD-1 or PDL-1 inhibitor. The single agent chemotherapy chosen is at the discretion of the site investigator and may include pemetrexed, gemcitabine or taxotere. Institutional standards should be used for administration of the single agent chemotherapy. For both treatment arms, 21 days equals 1 cycle of therapy and subjects will be eligible to continue treatment until progressive disease by RECIST v1.1 or unacceptable toxicity.

Upon registration, subjects will be randomized in a 1:1 ratio to either treatment with single agent chemotherapy or single agent chemotherapy in combination with nivolumab. Randomization is un-blinded and open-label; therefore there will be no placebo treatment for subjects randomized to single agent chemotherapy

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0-2 within 28 days prior to randomization.
4. Histological or cytological confirmed squamous or non-squamous non-small cell lung cancer.
5. Measurable disease according to RECIST 1.1 within 28 days prior to randomization.
6. A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to randomization, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic.
7. Subjects must have primary resistance to PD-1 or PDL-1 inhibitors; defined as PD after 3 or fewer treatments with a PD-1 or PDL-1 inhibitor
8. Subjects must have progressed on or after previous platinum-based chemotherapy. Chemotherapy may have previously been given with a PD-1 or PD-L1 inhibitor. Subjects must have also progressed on or after receiving any PD-1 or PD-L1 inhibitor (including nivolumab) as their most recent therapy.
9. Most recent PD-1 or PD-L1 inhibitor infusion must be completed at least 6 weeks of randomization. The subject must have recovered from all reversible acute toxic effects (other than alopecia) to ≤ Grade 1 or baseline.
10. Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to randomization.

    White blood cell (WBC) ≥ 2 k/mm3 Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3 Hemoglobin (Hgb) ≥ 9 g/dL Platelet >100k Estimated creatinine clearance OR ≥ 40 cc/min Serum creatinine ≤ 1.5 x upper limit of normal (ULN) Bilirubin 1.5 ≤ (ULN)2 Aspartate aminotransferase (AST) ≤ 1.5 × ULN Alanine aminotransferase (ALT) ≤ 1.5 × ULN International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤ 2 × ULN (Note: use of vitamin K antagonist is not allowed)
11. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days prior to registration. These women must also have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Nivolumab then every 6 weeks thereafter. NOTE: Women are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are post-menopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
12. Women of childbearing potential must be willing to abstain from heterosexual activity or use an effective method of contraception from the time of informed consent until 5 months after treatment discontinuation. Women cannot breast feed from the time of informed consent to 5 months after last dose of study treatment. See below for adequate methods of contraception.
13. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving Nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. See below for methods of contraception.
14. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria

1. Prior treatment with the single agent chemotherapy the site investigator chooses to use for this protocol (pemetrexed, taxotere or gemcitabine).
2. Previous autoimmune complication from PD-1 or PD-L1 requiring discontinuation of therapy or treatment with steroids (ongoing treatment with more than 10 mg of prednisone or steroid equivalent daily, excluding inhaled or topical steroids).
3. Previous discontinuation from PD-1 or PD-L1 due to an adverse event.
4. Any serious or uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy.
5. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
6. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
7. Active central nervous system (CNS) metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is 4 weeks or more] after treatment is complete and within 28 days prior to the first dose of Nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
8. Treatment with any investigational drug within 30 days prior to registration.
9. Subjects whose tumors express EGFR mutations on exons 19 and 21, ALK rearrangement, or ROS1 rearrangement who still have other FDA approved targeted agents available for treatment.
10. Subjects with an active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids/immunosuppressive medications EXCEPT for syndromes which would not be expected to recur in the absence of an external trigger. (Subjects with vitiligo, autoimmune thyroiditis, or type I diabetes mellitus are permitted to enroll.)
11. As there is potential for hepatic toxicity with Nivolumab, drugs with a predisposition to hepatoxicity should be used with caution in subjects treated with Nivolumab-containing regimen.
12. Subjects should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
13. Subjects should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
14. History of allergy to study drug components.
15. Prior solid organ or stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Principal Investigator — Hoosier Cancer Research Network
Locations (9):
- United States (9):
  - St. Vincent Anderson Regional Hospital, Anderson, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - IU Health Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - Community Healthcare System, Munster, Indiana
  - HealthPartners Institute, Minneapolis, Minnesota
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — https://hoosiercancer.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Single Agent Chemotherapy + Nivolumab: Single Agent Chemotherapy of choice plus nivolumab:
  Taxotere Pemetrexed Gemcitabine
  Docetaxel: Docetaxel 75 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
  Nivolumab: Nivolumab 360 mg IV Day 1 of each cycle (21 days = 1 cycle)
  Gemcitabine: Gemcitabine 1000 mg/m2 IV Day 1 and Day 8 of each cycle (21 days = 1 cycle)
  Pemetrexed: Pemetrexed 500 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
Period: Overall Study
Arm/Group | Arm A - Single Agent Chemotherapy + Nivolumab | Arm B - Single Agent Chemotherapy
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Disease Progression | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Single Agent Chemotherapy of choice plus nivolumab:
  Taxotere Pemetrexed Gemcitabine
  Docetaxel: Docetaxel 75 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
  Nivolumab: Nivolumab 360 mg IV Day 1 of each cycle (21 days = 1 cycle)
  Gemcitabine: Gemcitabine 1000 mg/m2 IV Day 1 and Day 8 of each cycle (21 days = 1 cycle)
  Pemetrexed: Pemetrexed 500 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
- Arm B: Single Agent Chemotherapy of choice Taxotere Pemetrexed Gemcitabine
  Docetaxel: Docetaxel 75 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
  Gemcitabine: Gemcitabine 1000 mg/m2 IV Day 1 and Day 8 of each cycle (21 days = 1 cycle)
  Pemetrexed: Pemetrexed 500 mg/m2 IV Day 1 of each cycle (21 days = 1 cycle)
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 1 | 2 | 3
  Large Cell Carcinoma | 0 | 0 | 0
  Mixed Histology | 0 | 0 | 0
  Non-small Cell Carcinoma | 0 | 0 | 0
  Sqamous | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS), as Defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Description: Compare PFS rates for subjects on each treatment arm, per RECIST 1.1. Subjects who have not progressed will be right-censored at the date of the last follow up.
Time Frame: 24 months
Population: Data for this objective was neither collected or analyzed due to the early termination of the study.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR) for Subjects on Each Treatment Arm, as Defined by RECIST 1.1 and Immune-related Response Criteria (irRECIST)
Description: Proportion of subjects on each arm with complete response or partial response, per RECIST 1.1 and irRECIST
Time Frame: Every 6 weeks beginning with C3D1 and every odd numbered cycle thereafter, assessed for up to 24 months
Population: Data for this objective was neither collected or analyzed due to the early termination of the study.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Clinical Benefit Rate (CBR) for Subjects on Each Treatment Arm, as Defined by RECIST 1.1 and irRECIST
Description: Proportion of subjects on each arm with complete response, partial response or stable disease for at least 3 months, per RECIST 1.1 and irRECIST
Time Frame: From D1 of treatment until documented disease progression/recurrence, assessed for up to 24 months
Population: Data for this objective was neither collected or analyzed due to the early termination of the study.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression Free Survival (PFS), as Defined by irRECIST
Description: Compare PFS rates for subjects on each treatment arm, per irRECIST. From date of randomization until the criteria for disease progression is met or death as a result of any cause, assessed up to 24 months
Time Frame: 24 months
Population: Data for this objective was neither collected or analyzed due to the early termination of the study.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Grade 3 or Grade 4 Adverse Events
Description: Assess toxicity of Nivolumab plus single agent chemotherapy compared with single agent chemotherapy alone. Number of grade 3 and 4 toxicities as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 1 | 2
participants
  GR4 Thromboembolic Event | 0 | 1
  GR3 Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are to be collected for the duration of the subject's participation on study, up to a maximum of six months.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=1) | Arm B (N=2)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=1) | Arm B (N=2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (2) | 0 (0)
HOT FLASHES (Vascular disorders) | 1 (1) | 0 (0)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 (2) | 0 (0)
LUNG INFECTION (Infections and infestations) | 1 (1) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to lack of accrual. Sufficient data was not collected to analyze any pre-specified endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT03041181/Prot_SAP_000.pdf